CLINICAL TRIAL: NCT01374373
Title: A Phase 4 Study in the Treatment of Anemia With Weekly Epoetin Alfa Doses in Patients With Solid Tumors or Lymphoma Receiving Chemotherapy
Brief Title: Epoetin Alfa (Hemax®) Phase IV Study in Chemotherapy Induced Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bio Sidus SA (Industry)
Collaborators: IC RESEARCH GROUP (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOS-012010
Record Dates: First submitted 2011-06-13; First posted 2011-06-16 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Antineoplastic Chemotherapy Induced Anemia
Keywords: Chemotherapy; Anemia; Epoetin alfa; Erythropoiesis stimulating agent (ESA)
MeSH Terms: conditions — Anemia | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label (Other): One arm open label
  Interventions: Biological: Epoetin alfa

INTERVENTIONS:
Biological: Epoetin alfa — Epoetin alfa 40.000-60.000 IU/week subcutaneously that will be controlled and up or down titrated every 2 weeks according to the currently approved prescription guidance for a total of 12 weeks of treatment with Co administration of oral ferrous sulfate 200mg BID and oral folic acid 5mg QD

SUMMARY:
The purpose of this study is to assess safety and efficacy of weekly epoetin alfa (Hemax® ) administered for 12 weeks in patients with non curable solid tumors or lymphoma with anemia (hemoglobin < 10g/dl) undergoing palliative care chemotherapy.

DETAILED DESCRIPTION:
Patients with non curable solid tumors or lymphoma with anemia (hemoglobin < 10g/dl) undergoing palliative care chemotherapy will enter this 12 week single arm open label study. Epoetin alfa 40.000-60.000 IU/week will be administered subcutaneously and controlled every 2 weeks. Up or down titration will be performed according to the currently approved prescription guidance for a total of 12 weeks of treatment. Study end points will be assessed every 4 weeks until final 12 week visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of non curable cancer or lymphoma
* Receiving a palliative chemotherapy regimen
* Hemoglobin < 10.0 g/dL
* Performance ≤ 3 of Eastern Cooperative Oncology Group (ECOG) performance status
* Life expectancy of ≥ 3 months
* Postmenopausal o premenopausal women receiving effective contraceptive method

Exclusion Criteria:

* Active bleeding that may have caused anemia in the prior 30 days.
* Uncontrolled hypertension
* Anemia for another cause other than cancer or chemotherapy
* Untreated iron or folic acid deficiency
* Transfusion in the last 30 days prior to baseline visit
* Treatment with an erythropoiesis stimulating agent 3 months prior to the baseline visit
* Increased risk of thromboembolic disease
* Radiotherapy in pelvis or spine in the last 60 days
* Myelodysplasic syndrome
* History of congestive heart failure
* Pregnant or lactating
* Patient with known allergy to human albumin or related products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and percentage of therapy withdrawals due to treatment emergent adverse events | Baseline to 12 weeks

SECONDARY OUTCOMES:
Hemoglobin levels and percentage of responders | Every 4 weeks and 12 weeks
  Evaluate efficacy assessing hemoglobin levels and percentage of responders (increments of Hemoglobin ≥ 1g/dl without transfusion requirements) comparing baseline with final 12 week and intermediate 4 week visits
Quality of life | 12 Weeks
  Evaluate if treatment impacts quality of life assessed through the Brief Fatigue Index (BFI) score comparing baseline with final 12 week visit
Hemoglobin levels ≥ 2 g/dl | 12 weeks
  Evaluate proportion of patient that achieve hemoglobin levels ≥ 2 g/dl without transfusion requirements and the number of patients that require at least one transfusion after 12 weeks of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Diez, MD, Study Director — Bio Sidus SA
Locations (3):
- Argentina (3):
  - Centro Oncologico de Investigaciones Buenos Aires, Berazategui, Buenos Aires
  - Centro de Medicina Integral e Investigación Clínica, Buenos Aires, Buenos Aires
  - Hospital Zonal Especializado en Oncología de Lanus, Lanús Este, Buenos Aires